CLINICAL TRIAL: NCT06244082
Title: A Phase 2 Open-label Study to Evaluate the Pharmacodynamics and Long-Term Safety and Tolerability of AOC 1044 Administered Intravenously to DMD Participants With Mutations Amenable to Exon 44 Skipping
Brief Title: Ph2 Open-label Study of AOC 1044 in Duchenne Muscular Dystrophy Participants With Mutations Amenable to Exon44 Skipping
Acronym: EXPLORE44OLE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Avidity Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOC 1044-CS2
Record Dates: First submitted 2024-01-26; First posted 2024-02-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: DMD; Duchenne Muscular Dystrophy; Duchenne; Exon 44
Keywords: EXPLORE44; EXPLORE44-OLE; EXPLORE44 OLE; Avidity Biosciences; Avidity; AOC 1044; AOC 1044-CS1; AOC 1044-CS2; AOC
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Masking Description: Randomization from the parent study, AOC 1044-CS1 will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AOC 1044 Multiple Dose Levels (Experimental): AOC 1044 will be IV infused every 6 weeks for approximately 2 years.
  Interventions: Drug: AOC 1044

INTERVENTIONS:
Drug: AOC 1044 — AOC 1044 will be administered via intravenous (IV) infusion

SUMMARY:
AOC 1044-CS2 (EXPLORE44-OLE) is an Open-label Study to Evaluate the Long-Term Safety and Tolerability of AOC 1044 Administered Intravenously to DMD Participants with Mutations Amenable to Exon 44 Skipping.

DETAILED DESCRIPTION:
AOC 1044-CS2 (EXPLORE44-OLE) is an open label, extension study to Part B of AOC 1044-CS1 (EXPLORE44). AOC 1044-CS2 is designed to evaluate the long-term safety, tolerability, pharmacokinetics, and exploratory efficacy of AOC 1044.

All participants who enroll in AOC 1044-CS2 will receive active treatment. The treatment period is 2 years with IV dosing every 6 weeks.

Once participants have completed active treatment, they will be followed through a 3-month safety follow-up period. The sponsor may extend active treatment beyond 2 years at a future timepoint.

ELIGIBILITY:
Key Inclusion Criteria

Rollover Participants:

* Satisfactorily completed AOC 1044-CS1 (EXPLORE44) as determined by the Investigator and Sponsor
* No significant tolerability issues with AOC 1044

De novo Participants:

* Aged 7 to 27 years, inclusive, at the time of informed consent
* Clinical diagnosis of DMD or clear onset of DMD symptoms at or before the age of 6 years
* Confirmation of DMD gene mutation amenable to exon 44 skipping
* Weight ≥ 23 kg
* Ambulatory or non-ambulatory

  * Ambulatory participants: LVEF ≥50% and FVC≥50%
  * Non-ambulatory participants: LVEF ≥45% and FVC≥40%
* PUL 2.0 entry item A ≥3
* If on corticosteroids, stable dose for 30 days before screening and throughout the study

Key Exclusion Criteria

Rollover Participants:

* Presence of any new condition or worsening of existing condition that could affect a participant's safety or ability to comply with study procedures

De novo Participants:

* Serum hemoglobin < lower limit of normal
* Uncontrolled hypertension or diabetes
* Prior treatment with any cell or gene therapy
* Prior treatment with another exon 44 skipping agent within 6 months prior to informed consent
* Recently treated with an investigational drug
* History of multiple drug allergies

Ages: 7 Years to 27 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Through study completion (approximately 2 years)

SECONDARY OUTCOMES:
Change from baseline in serum creatine kinase concentration at Study Weeks 24, 48, and 102 | Through study completion (approximately 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Castrillo, MD, Study Director — Avidity Biosciences, Inc.
Locations (10):
- United States (10):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California, San Diego, Rady's Children's Hospital, La Jolla, California
  - UC Davis Medical Center, Sacramento, California
  - Lucille Packard Children's Hospital at Stanford, San Carlos, California
  - Rare Disease Research - Atlanta, Atlanta, Georgia
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Rare Disease Research, Hillsborough, North Carolina
  - Abigail Wexner Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Neurology Rare Disease Center, Denton, Texas

IPD SHARING:
Plan to Share IPD: No